CLINICAL TRIAL: NCT00074386
Title: Solid Organ Transplantation in HIV: Multi-Site Study
Brief Title: Kidney and Liver Transplantation in People With HIV
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1U01AI052748 (NIH); 1U01AI052748 (NIH); NCT00023478 (obsolete NCT alias); NCT00473629 (obsolete NCT alias)
Record Dates: First submitted 2003-12-11; First posted 2003-12-15 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections; Kidney Disease; Liver Disease
Keywords: HIV; Transplant; Liver; Kidney; Organ; Treatment Experienced; Kidney Transplant; Liver Transplant
MeSH Terms: conditions — HIV Infections; Kidney Diseases; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, serum, PBMC, kidney and liver biopsy slides, saliva, spleen tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With improved anti-HIV drug therapy, HIV infected patients are now living longer. These patients are at risk for liver and kidney failure and may need organ transplants. However, little is know about the safety and effectiveness of organ transplants in patients with HIV. This study will evaluate organ transplantation in HIV infected patients undergoing liver and kidney transplants.

DETAILED DESCRIPTION:
HIV infected people are at significant risk for end stage organ disease. Prior to the advent of highly active antiretroviral therapy (HAART), these people were often not considered transplant candidates based on concern about potential adverse effects of immunosuppressive drugs on HIV disease progression. However, with the use of HAART, HIV infected people have experienced significant improvements in morbidity and mortality. HIV infected people with end stage kidney and liver disease are now potential candidates for transplantation, yet patients and clinicians lack the necessary data to determine the safety and efficacy of transplantation and immunosuppression in this group. This lack of conclusive data has led to continued denial of care by many transplant centers and third party payers, resulting in frustration and confusion for both patients and their health care providers.

This study will evaluate the safety and efficacy of solid organ transplantation in people with HIV infection by following a prospective, multi-center cohort of HIV infected people who undergo kidney or liver transplantation. The long-term goals are: 1) to provide patients and clinicians with information regarding the HIV-specific risks of transplantation; 2) to provide clinicians with information necessary to manage immunosuppressive and HAART medications together; and 3) to understand underlying basic science mechanisms that explain patient outcomes so that clinical management can be adjusted to improve outcomes.

Approximately 150 kidney and 125 liver transplant patients will be enrolled in this study over a 3-year period at medical research centers throughout the United States. Participants will be enrolled in the study for five years from the day of the transplant.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infection
* Undetectable HIV viral load
* Meet all eligibility requirements for a transplant (same requirements that HIV uninfected patients must meet)
* Willing to take medication to prevent certain infections
* Willing to undergo frequent monitoring, including liver biopsies, and treatment, if participant has hepatitis B or C virus infection
* Willing to submit laboratory test results within 7 days of blood draw
* Willing to notify the transplant team before changing any medications
* If participant has a history of HIV-related cancers or opportunistic infections, some additional eligibility criteria must be met.

Inclusion Criteria for Patients Undergoing Kidney Transplant:

* CD4 count greater than 200 cells/mm3. CD4 count requirement for children will be based on child's age. Participant cannot have used the drugs IL-2 or GM-CSF in order to increase the CD4 count in the 6 months prior to transplant.

Inclusion Criteria for Patients Undergoing Liver Transplant:

* CD4 count greater than 100 cells/mm3. CD4 count requirement for children will be based on child's age. Some participants with certain HIV-related diseases must have a CD4 count that is greater than 200 cells/ml for the 6 months prior to study entry.

Exclusion Criteria for All Participants:

* Pregnancy
* Significant wasting or weight loss

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-positive patients who undergo kidney or liver transplantation.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2003-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Subject survival | 5 years
graft survival | 5 years

SECONDARY OUTCOMES:
Opportunistic complications | 5 years
CD4+ T cell counts and HIV-1 RNA levels | 5 years
viral markers and host-response (CFC and ELISPOT) to viral co-pathogens, including HBV, HCV,CMV, EBV, HHV-6, HHV-8, and HPV | 5 years
rejection rates and markers of alloresponse | 5 years
pharmacokinetic interactions between immunosuppressive agents and antiretrovirals | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stock, MD, Principal Investigator — University of California, San Francisco; Michelle Roland, Principal Investigator — University of California, San Francisco
Locations (21):
- United States (21):
  - Cedar-Sinai Hospital, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami, Jackson Memorial Medical Center, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess, Boston, Massachusetts
  - Mt. Sinai Medical Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - The University Hospital, Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Thomas E. Starzl Institute, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Terrault NA, Roland ME, Schiano T, Dove L, Wong MT, Poordad F, Ragni MV, Barin B, Simon D, Olthoff KM, Johnson L, Stosor V, Jayaweera D, Fung J, Sherman KE, Subramanian A, Millis JM, Slakey D, Berg CL, Carlson L, Ferrell L, Stablein DM, Odim J, Fox L, Stock PG; Solid Organ Transplantation in HIV: Multi-Site Study Investigators. Outcomes of liver transplant recipients with hepatitis C and human immunodeficiency virus coinfection. Liver Transpl. 2012 Jun;18(6):716-26. doi: 10.1002/lt.23411. PMID 22328294
- [Result] Carter JT, Melcher ML, Carlson LL, Roland ME, Stock PG. Thymoglobulin-associated Cd4+ T-cell depletion and infection risk in HIV-infected renal transplant recipients. Am J Transplant. 2006 Apr;6(4):753-60. doi: 10.1111/j.1600-6143.2006.01238.x. PMID 16539632
- [Result] Frassetto L, Baluom M, Jacobsen W, Christians U, Roland ME, Stock PG, Carlson L, Benet LZ. Cyclosporine pharmacokinetics and dosing modifications in human immunodeficiency virus-infected liver and kidney transplant recipients. Transplantation. 2005 Jul 15;80(1):13-7. doi: 10.1097/01.tp.0000165111.09687.4e. PMID 16003227
- [Result] Roland ME, Carlson LL, Frassetto LA, Stock PG. Solid organ transplantation: referral, management, and outcomes in HIV-infected patients. AIDS Read. 2006 Dec;16(12):664-8, 675-8. PMID 17195325
- [Result] Roland ME, Stock PG. Liver transplantation in HIV-infected recipients. Semin Liver Dis. 2006 Aug;26(3):273-84. doi: 10.1055/s-2006-947297. PMID 16850377
- [Result] Roland ME, Stock PG. Solid organ transplantation is a reality for patients with HIV infection. Curr HIV/AIDS Rep. 2006 Sep;3(3):132-8. doi: 10.1007/BF02696657. PMID 16970840
- [Result] Terrault NA, Carter JT, Carlson L, Roland ME, Stock PG. Outcome of patients with hepatitis B virus and human immunodeficiency virus infections referred for liver transplantation. Liver Transpl. 2006 May;12(5):801-7. doi: 10.1002/lt.20776. PMID 16628690
- [Result] Bihl FK, Loggi E, Chisholm JV 3rd, Hewitt HS, Henry LM, Linde C, Suscovich TJ, Wong JT, Frahm N, Andreone P, Brander C. Simultaneous assessment of cytotoxic T lymphocyte responses against multiple viral infections by combined usage of optimal epitope matrices, anti- CD3 mAb T-cell expansion and "RecycleSpot". J Transl Med. 2005 May 11;3(1):20. doi: 10.1186/1479-5876-3-20. PMID 15888204
- [Result] Frassetto LA, Browne M, Cheng A, Wolfe AR, Roland ME, Stock PG, Carlson L, Benet LZ. Immunosuppressant pharmacokinetics and dosing modifications in HIV-1 infected liver and kidney transplant recipients. Am J Transplant. 2007 Dec;7(12):2816-20. doi: 10.1111/j.1600-6143.2007.02007.x. Epub 2007 Oct 19. PMID 17949460
- [Result] Stock PG, Roland ME. Evolving clinical strategies for transplantation in the HIV-positive recipient. Transplantation. 2007 Sep 15;84(5):563-71. doi: 10.1097/01.tp.0000279190.96029.77. PMID 17876267
- [Result] Frassetto LA, Tan-Tam C, Stock PG. Renal transplantation in patients with HIV. Nat Rev Nephrol. 2009 Oct;5(10):582-9. doi: 10.1038/nrneph.2009.140. PMID 19776780
- [Result] Subramanian A, Sulkowski M, Barin B, Stablein D, Curry M, Nissen N, Dove L, Roland M, Florman S, Blumberg E, Stosor V, Jayaweera DT, Huprikar S, Fung J, Pruett T, Stock P, Ragni M. MELD score is an important predictor of pretransplantation mortality in HIV-infected liver transplant candidates. Gastroenterology. 2010 Jan;138(1):159-64. doi: 10.1053/j.gastro.2009.09.053. Epub 2009 Sep 30. PMID 19800334
- [Result] Gasser O, Bihl F, Sanghavi S, Rinaldo C, Rowe D, Hess C, Stablein D, Roland M, Stock P, Brander C. Treatment-dependent loss of polyfunctional CD8+ T-cell responses in HIV-infected kidney transplant recipients is associated with herpesvirus reactivation. Am J Transplant. 2009 Apr;9(4):794-803. doi: 10.1111/j.1600-6143.2008.02539.x. PMID 19298451
- [Result] Coffin CS, Stock PG, Dove LM, Berg CL, Nissen NN, Curry MP, Ragni M, Regenstein FG, Sherman KE, Roland ME, Terrault NA. Virologic and clinical outcomes of hepatitis B virus infection in HIV-HBV coinfected transplant recipients. Am J Transplant. 2010 May;10(5):1268-75. doi: 10.1111/j.1600-6143.2010.03070.x. Epub 2010 Mar 19. PMID 20346065
- [Result] Tan-Tam CC, Frassetto LA, Stock PG. Liver and kidney transplantation in HIV-infected patients. AIDS Rev. 2009 Oct-Dec;11(4):190-204. PMID 19940946
- [Result] Stock PG, Barin B, Murphy B, Hanto D, Diego JM, Light J, Davis C, Blumberg E, Simon D, Subramanian A, Millis JM, Lyon GM, Brayman K, Slakey D, Shapiro R, Melancon J, Jacobson JM, Stosor V, Olson JL, Stablein DM, Roland ME. Outcomes of kidney transplantation in HIV-infected recipients. N Engl J Med. 2010 Nov 18;363(21):2004-14. doi: 10.1056/NEJMoa1001197. PMID 21083386
- [Result] Harbell J, Fung J, Nissen N, Olthoff K, Florman SS, Hanto DW, Light J, Bartlett ST, Tzakis AG, Pearson TC, Barin B, Roland ME, Stock PG; HIV-TR Investigators. Surgical complications in 275 HIV-infected liver and/or kidney transplantation recipients. Surgery. 2012 Sep;152(3):376-81. doi: 10.1016/j.surg.2012.06.012. PMID 22938898
- [Result] Nissen NN, Barin B, Stock PG. Malignancy in the HIV-infected patients undergoing liver and kidney transplantation. Curr Opin Oncol. 2012 Sep;24(5):517-21. doi: 10.1097/CCO.0b013e328355e0d7. PMID 22759736
- [Result] Ragni MV, Devera ME, Roland ME, Wong M, Stosor V, Sherman KE, Hardy D, Blumberg E, Fung J, Barin B, Stablein D, Stock PG. Liver transplant outcomes in HIV+ haemophilic men. Haemophilia. 2013 Jan;19(1):134-40. doi: 10.1111/j.1365-2516.2012.02905.x. Epub 2012 Jul 5. PMID 22762561
- [Result] Ansari IU, Allen T, Berical A, Stock PG, Barin B, Striker R. Phenotypic analysis of NS5A variant from liver transplant patient with increased cyclosporine susceptibility. Virology. 2013 Feb 20;436(2):268-73. doi: 10.1016/j.virol.2012.11.018. Epub 2013 Jan 2. PMID 23290631
- [Result] Bahirwani R, Barin B, Olthoff K, Stock P, Murphy B, Rajender Reddy K; Solid Organ Transplantation in HIV: Multi-Site Study Investigators. Chronic kidney disease after liver transplantation in human immunodeficiency virus/hepatitis C virus-coinfected recipients versus human immunodeficiency virus-infected recipients without hepatitis C virus: results from the National Institutes of Health multi-site study. Liver Transpl. 2013 Jun;19(6):619-26. doi: 10.1002/lt.23648. PMID 23512786
- [Result] Chin-Hong P, Beatty G, Stock P. Perspectives on liver and kidney transplantation in the human immunodeficiency virus-infected patient. Infect Dis Clin North Am. 2013 Jun;27(2):459-71. doi: 10.1016/j.idc.2013.02.010. Epub 2013 Mar 29. PMID 23714349
- [Result] Frassetto L, Floren L, Barin B, Browne M, Wolfe A, Roland M, Stock P, Carlson L, Christians U, Benet L. Changes in clearance, volume and bioavailability of immunosuppressants when given with HAART in HIV-1 infected liver and kidney transplant recipients. Biopharm Drug Dispos. 2013 Nov;34(8):442-51. doi: 10.1002/bdd.1860. Epub 2013 Sep 12. PMID 24030928
- [Result] Gregg KS, Barin B, Pitrak D, Ramaprasad C, Pursell K. Acquired hypogammaglobulinemia in HIV-positive subjects after liver transplantation. Transpl Infect Dis. 2013 Dec;15(6):581-7. doi: 10.1111/tid.12139. Epub 2013 Sep 18. PMID 24103022
- [Derived] Roland ME, Barin B, Huprikar S, Murphy B, Hanto DW, Blumberg E, Olthoff K, Simon D, Hardy WD, Beatty G, Stock PG; HIVTR Study Team. Survival in HIV-positive transplant recipients compared with transplant candidates and with HIV-negative controls. AIDS. 2016 Jan 28;30(3):435-44. doi: 10.1097/QAD.0000000000000934. PMID 26765937
- [Derived] Stock PG, Terrault NA. Human immunodeficiency virus and liver transplantation: Hepatitis C is the last hurdle. Hepatology. 2015 May;61(5):1747-54. doi: 10.1002/hep.27553. Epub 2015 Mar 19. No abstract available. PMID 25292153
- [Derived] Sherman KE, Terrault N, Barin B, Rouster SD, Shata MT; HIV-TR Investigators. Hepatitis E infection in HIV-infected liver and kidney transplant candidates. J Viral Hepat. 2014 Aug;21(8):e74-7. doi: 10.1111/jvh.12233. Epub 2014 Apr 28. PMID 24773782
- [Derived] Frassetto LA, Tan-Tam CC, Barin B, Browne M, Wolfe AR, Stock PG, Roland M, Benet LZ. Best single time point correlations with AUC for cyclosporine and tacrolimus in HIV-infected kidney and liver transplant recipients. Transplantation. 2014 Mar 27;97(6):702-7. doi: 10.1097/01.TP.0000441097.30094.31. PMID 24389906